## **Statistical Analysis Plan**

Title: Ultrasound-guided Intermediate Cervical Plexus Block

ID A 2016 0027 NCT 02794974

The metric parameters are described by mean value (Mw) and standard deviation (Sd). The Mann-Whitney U test tests whether the two groups differ in the distribution of the parameter. If the p-value of the test is less than the selected significance level (0.05), then the groups differ significantly in terms of distribution.

Categorical parameters (0/1) are described by the exact Fisher test. The exact Fisher test examines whether each parameter is independent of its membership in a group. If the p-value of the test is less than the selected significance level (0.05), then there is a significant dependence. The two groups then differ significantly with respect to the selected parameter.

The incidence of adverse events in the two groups is described with odds ratios (95% confidence interval).

All statistical tests were performed bilaterally at significance level 0.05. Stata 14.2 / IC for Windows was used for the statistical analysis. All tests were carried out by a professional statistician (www.p-wert.de).